CLINICAL TRIAL: NCT06443034
Title: Predictive Determinants of Nephrotic Syndrome Remission in Patients With Focal Segmental Glomerulosclerosis or Minimal Change Disease and At-risk Polymorphism of APOL1 Gene
Brief Title: Predictive Determinants of Nephrotic Syndrome Remission in Patients With At-risk Polymorphism of APOL1
Acronym: NEPHROL1
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240269
Record Dates: First submitted 2024-05-28; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Nephrotic Syndrome; Focal Segmental Glomerulosclerosis; APOL1 Associated Kidney Disease
Keywords: Nephrotic syndrome; Covid-19 associated nephropathy; human immunodeficiency virus associated nephropathy; APOL1 associated kidney disease; Focal segmental glomerulosclerosis; Minimal change disease
MeSH Terms: conditions — Nephrotic Syndrome; Glomerulosclerosis, Focal Segmental; AIDS-Associated Nephropathy; Nephrosis, Lipoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicentric retrospective observational cohort study.

As primary objective, the study aims to evaluate the factors associated with nephrotic syndrome remission in patient with nephrotic syndrome, biopsy-prove minimal change disease or focal segmental glomerulosclerosis, and an at-risk variant of the APOL1 gene.

As secondary objectives, this study aims:

* To evaluate the benefit of corticosteroids in obtaining the remission of nephrotic syndrome
* To identify the predictors of complete renal remission of nephrotic syndrome
* To evaluate the benefit of corticosteroids in reducing the incidence of end-stage renal disease
* To assess the adverse events of corticosteroids in patients treated with corticosteroids.

DETAILED DESCRIPTION:
The APOL1 gene synthesizes Apolipoprotein L1, a transport protein for hydrophobic molecules. When this gene presents bi-allelic "at risk" polymorphisms, it has been associated with an increased risk of end-stage renal disease. These polymorphisms can be frequent on a population scale, affecting up to 32% of patients in some West African countries. The pathogenic nature of these variants is now well established and has been highlighted on several occasions, notably in HIV-associated nephropathy (HIVAN - HIV Associated Nephropathy) or more recently in COVID-19-associated nephropathy (COVAN - COVID Associated Nephropathy), where almost all patients carry APOL1 risk alleles. Irrespective of the causative agent, nephropathy associated with APOL1 risk variants is regularly revealed by a nephrotic syndrome. This syndrome is characterized by generalized edema, high-range proteinuria and acute kidney injury. The course of the disease is particularly difficult to predict and highly variable, with some patients requiring rapid and definitive dialysis while others recover normal renal function without sequelae of proteinuria. In addition to this inter-individual variability, there is also variability in clinical practice with regard to the use of high-dose corticosteroids to induce disease remission. This is largely due to the rarity of the disease in the West and its possible under-diagnosis in developing countries. However, new drugs specifically targeting APOL1 are currently being developed, but their use is currently restricted to studies that exclude the most severe patients. In patients with at-risk APOL1 variants and nephrotic syndromes, it therefore appears critical to identify the determinants associated with remission of nephropathy, to quantify the efficacy of current therapies and to facilitate access to emerging drugs for the most severely ill subjects.

The main aim of this study is to evaluate the predictors (drug, clinical, histological or biological parameters) associated with nephrotic syndrome remission in patients with nephrotic syndrome, biopsy proven focal segmental glomerulosclerosis or minimal change disease and an at-risk variant of the APOL1 gene.

Population involved: eligible patients will be enrolled if they are more than 18 years old, have nephrotic syndrome (serum albumin < 30 g/L and urine protein creatinine ratio > 3 g/g) and biopsy-proven focal segmental glomerulosclerosis or minimal change disease.

Data analysis: the association of each explanatory variable with the variable "remission of nephrotic syndrome" will first be assessed using a semi-parametric univariable Cox model.Then, a multivariable Cox model will be performed with the explanatory variables associated with the variable "remission of nephrotic syndrome" with a p value < 0.2 at the Wald test in univariable Cox regression analysis. Variables independently associated with remission of nephrotic syndrome will be those with a two-sided p value < 0.05 after stepwise backward elimination in the multivariate model.

In order to assess the robustness of our results with the statistical approach, the investigators will also conduct association analyses between the predictor variables and the variable of interest using the machine learning analysis known as "Random Forrest analysis".

As secondary outcomes, the association between corticosteroids and nephrotic syndrome remission will be evaluated. The association between corticosteroids and end-stage renal disease will also be evaluated as a secondary outcome. The third secondary outcome evaluated will be the association between the predictor variables and complete remission of nephrotic syndrome. The last secondary outcome will be the assessment of corticosteroids safety evaluated following the common terminology criteria for adverse event version 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients followed in 6 nephrology centers between 01/01/2016 and 01/06/2024.
* With characterization of APOL1 gene risk status
* Proteinuria/creatinuria ratio > 3 g/g at diagnosis of renal disease (within 48 hours of the diagnostic renal biopsy)
* Hypoalbuminemia < 30 g/L at diagnosis of renal disease (within 48 h of diagnostic renal biopsy)
* Minimal change disease or segmental and focal hyalinosis lesions on renal biopsy.

Exclusion Criteria:

* Presence of diffuse deposits of immunoglobulins or complement fractions on immunofluorescence study
* Presence of endo- or extracapillary hypercellular lesions on light microscopy
* Opposition to the use of medical data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients APOL1 gene status will be obtained from the Hôpital Européen Georges Pompidou genetic laboratory (performing all APOL1 gene analysis in Paris greater area).
  Patients with a biopsy-proven focal segmental glomerulosclerosis or minimal change disease and nephrotic syndrome will be screened in each center.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
nephrotic syndrome remission | up to 12 months
  Description: remission of nephrotic syndrome is defined as a complete or partial remission of nephrotic syndrome as follows:
  * Complete remission:
    * Urine protein / creatinine ratio < 0.3 g/g AND
    * Albuminemia > 35 g/L
  * Partial remission:
    * Urine protein / creatinine ratio > 0.3 g/g AND
    * Urine protein / creatinine ratio < 3.5 g/g AND
    * > 50% reduction of urine protein / creatinine ratio from baseline (at the time of biopsy)

SECONDARY OUTCOMES:
end stage renal disease | up to 12 months
  estimated glomerular filtration rate (eGFR) below 15 ml/min/1.73m2 repeatedly over a period > 3 months OR dialysis > 3 months OR kidney transplantation.
complete remission of nephrotic syndrome Time Frame : between kidney biopsy and last follow-up | up to 12 months
  Urine protein / creatinine ratio < 0.3 g/g AND Albuminemia > 35 g/L
adverse effects of corticosteroids | up to 12 months
  The number of serious adverse events will be measured in patients treated with corticosteroids according to the CTCAE toxicity grading system for the following adverse events combined: death (all causes), grade 3 or higher infections, sickle cell disease vaso-occlusive crisis, and new-onset or hospitalization-requiring diabetes mellitus.

CONTACTS AND LOCATIONS:
Locations (1):
- Néphrologie & Dialyses department, Tenon Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided